CLINICAL TRIAL: NCT05968326
Title: A Phase II, Open-Label, Multicenter, Randomized Study of the Efficacy and Safety of Adjuvant Autogene Cevumeran Plus Atezolizumab and mFOLFIRINOX Versus mFOLFIRINOX Alone in Patients With Resected Pancreatic Ductal Adenocarcinoma
Brief Title: A Study of the Efficacy and Safety of Adjuvant Autogene Cevumeran Plus Atezolizumab and mFOLFIRINOX Versus mFOLFIRINOX Alone in Participants With Resected PDAC
Acronym: IMCODE003
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Collaborators: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO44479; 2022-502404-73-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2023-07-21; First posted 2023-08-01 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Adenocarcinoma, Pancreatic Ductal
MeSH Terms: conditions — Adenocarcinoma | interventions — atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: Autogene Cevumeran + Atezolizumab + mFOLFIRINOX (Experimental): Participants will receive autogene cevumeran, atezolizumab and mFOLFIRINOX.
  Interventions: Drug: Autogene cevumeran; Drug: Atezolizumab; Drug: mFOLFIRINOX
- Arm 2: mFOLFIRINOX (Active Comparator): Participants will receive mFOLFIRINOX.
  Interventions: Drug: mFOLFIRINOX

INTERVENTIONS:
Drug: Autogene cevumeran — Autogene cevumeran will be administered intravenously (IV) at a recommended dose at specified timepoints.
  Arms: Arm 1: Autogene Cevumeran + Atezolizumab + mFOLFIRINOX
Drug: Atezolizumab — Atezolizumab will be administered IV at a dose of 1680 milligrams (mg) at specified timepoints.
  Other Names: Tecentriq
  Arms: Arm 1: Autogene Cevumeran + Atezolizumab + mFOLFIRINOX
Drug: mFOLFIRINOX — mFOLFIRINOX (oxaliplatin, leucovorin, irinotecan, 5-FU) will be administered IV at specified timepoints.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of adjuvant autogene cevumeran plus atezolizumab and modified leucovorin, 5-fluorouracil (5-FU), irinotecan, and oxaliplatin (mFOLFIRINOX) versus mFOLFIRINOX alone in participants with resected pancreatic ductal adenocarcinoma (PDAC) who have not received prior systemic anti-cancer treatment for PDAC and have no evidence of disease after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of PDAC
* Pancreatic cancer tumor, lymph node, metastasis (TNM) pathological staging values of T1-T3, N0-N2, and M0 per the American Joint Committee on Cancer (AJCC) Cancer Staging Manual
* Macroscopically complete (R0 or R1) resection of PDAC
* Unequivocal absence of disease after surgery as assessed by the investigator within 28 days prior to treatment initiation
* CA19-9 level measured within 14 days prior to initiation of study treatment
* Interval of between 6 and 12 weeks since resection of PDAC
* Full recovery from surgery and ability to receive atezolizumab, autogene cevumeran, and mFOLFIRINOX in the investigator's judgment
* Adequate hematologic and end-organ function
* Female participants of childbearing potential must be willing to avoid pregnancy during the treatment period and for 28 days after the final dose of autogene cevumeran, for 9 months after the last dose of chemotherapy, and for 5 months after the final dose of atezolizumab. They must refrain from donating eggs for 9 months after the last dose of chemotherapy.
* Male participants with a female partner of childbearing potential or pregnant female partner must remain abstinent or use specified contraceptive methods during the treatment period and for 28 days after the final dose of autogene cevumeran and for 6 months after the last dose of chemotherapy. Men must refrain from donating sperm during this same period.

Exclusion Criteria:

* Prior adjuvant, neoadjuvant, or induction treatment for pancreatic cancer
* Plan for further adjuvant anti-cancer therapy for PDAC (e.g., radiotherapy and/or chemotherapy), not mandated per protocol, to be initiated after completion of mFOLFIRINOX treatment
* Absence of spleen; distal pancreatectomy with splenectomy is exclusionary
* Preexisting Grade >/=2 neuropathy
* Known complete dihydropyrimidine dehydrogenase (DPD) deficiency including homozygous or compound heterozygous mutations of DPYD genetic locus associated with DPD deficiency
* Disorders of the colon or rectum, or postoperative complication leading to Grade >/=2 diarrhea
* Pregnancy or breastfeeding
* Active or history of autoimmune disease or immune deficiency
* Treatment with brivudine, sorivudine, or their chemically-related analogues, which are inhibitors of DPD, within 4 weeks prior to initiation of study treatment
* Current or planned treatment with strong inhibitors or inducers of cytochrome P450 3A4 (CYP3A4) and/or uridine diphosphate glucoronosyltransferase 1A1 (UGT1A1).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2031-01-01 (Estimated); Study Completion 2031-01-01 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival (DFS) | From randomization to first recurrence of PDAC or first occurrence of new cancer, as determined by the investigator, or death from any cause (whichever occurs first), up to approximately 6 years

SECONDARY OUTCOMES:
DFS Rates at 12, 24, and 36 Months | Months 12, 24, 36
Overall Survival (OS) | From randomization to death from any cause (up to approximately 6 years)
OS Rates at 3 and 5 Years | Years 3 and 5
Percentage of Participants With Adverse Events (AEs) | Up to approximately 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (89):
- United States (32):
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - USC Norris Cancer Center, Newport Beach, California
  - University of California, San Francisco (UCSF), San Francisco, California
  - University of California Los Angeles, Santa Monica, California
  - St. Francis Hospital and Medical Center, Hartford, Connecticut
  - Smilow Cancer Center, New Haven, Connecticut
  - Yale Cancer Center, New Haven, Connecticut
  - Smilow Cancer Hospital Care Center at Trumbull, Trumbull, Connecticut
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Indiana University Health Melvin & Bren Simon Cancer Center, Indianapolis, Indiana
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Harvard Medical School - Massachusetts General Hospital (MGH) - Cancer Center, Boston, Massachusetts
  - Boston Medical Center (BMC) - Cancer Care Center, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - University of Nebraska, Omaha, Nebraska
  - Memorial Sloan Kettering Cancer Center Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center, Middletown, New Jersey
  - Memorial Sloan Kettering Cancer Center at Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center - Commack, Commack, New York
  - Memorial Sloan Kettering Cancer Center at Westchester, Harrison, New York
  - Northwell Health, Lake Success, New York
  - NYU Langone Health, New York, New York
  - Mount SInai Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - MEETH-LHH Northwell Health Cancer Clinical Trials Office at MEETH-LHH, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center at Nassau, Uniondale, New York
  - Duke Cancer Institute, Durham, North Carolina
  - University of Cincinnati Cancer Institute, Cincinnati, Ohio
  - Rhode Island Hospital, Providence, Rhode Island
  - Miriam Hospital, Providence, Rhode Island
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Belgium (5):
  - ULB Hôpital Erasme, Brussels
  - Antwerp University Hospital, Edegem
  - AZ Maria Middelares, Ghent
  - Universitair Ziekenhuis Gent, Ghent
  - UZ Leuven, Leuven
- Canada (4):
  - St Michael Hospital, Toronto, Ontario
  - Princess Margaret Cancer Center, Toronto, Ontario
  - Centre Hospitalier de l'Universite de Montreal - Notre - Dame Hos pital, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
- France (5):
  - Centre Hospitalier Régional Universitaire de Lille, Lille
  - Centre Leon Berard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif
- Germany (13):
  - Charite-Universitaetsmedizin Berlin - Campus Virchow-Klinikum (CVK), Berlin
  - Katholisches Klinikum Bochum gGmbH;St. Josef-Hospital, Bochum
  - Universitaetsklinikum Koeln, Cologne
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - Universitätsklinikum Essen, Essen
  - Krankenhaus Nordwest GmbH, Frankfurt
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Ludwig-Maximilians-Universität München, München
  - Klinikum Bogenhausen, München
  - Universitaetsklinikum Tuebingen, Tübingen
  - Universitätsklinikum Ulm, Klinik für Innere MedizinInnere Medizin III Studienzentrale, Ulm
  - Uniklinikum Würzburg, Med. Klinik und Poliklinik II, Würzburg
- Netherlands (3):
  - Amsterdam UMC Location VUMC, Amsterdam
  - UMC Radboud Nijmegen, Nijmegen
  - Erasmus MC, Rotterdam
- South Korea (7):
  - National Cancer Center (NCC) Hospital - Center for Liver and Pancreatobiliary Cancer, Goyang-si
  - CHA Bundang Medical Center, Gyeonggi-do
  - The Catholic University of Korea - Seoul St. Mary's Hospital (Kangnam St. Mary's Hospital), Seocho
  - Seoul National University Bundang Hospital, Seongnam-si
  - Samsung Medical Center, Seoul
  - Severance Hospital - Yonsei Cancer Center, Seoul
  - University of Ulsan College of Medicine - Asan Medical Center (AMC) - Asan Cancer Center (ACC), Songpa-gu
- Spain (10):
  - Institut Catala d?Oncologia Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Regional Universitario de Malaga, Málaga, Malaga
  - Clinica Universitaria de Navarra (CUN), Pamplona/iruña, Navarre
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario Vall d Hebron, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Clinica Universitaria de Navarra de Madrid;Servicio de Hepatologia, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario 12 De Octubre, Madrid
  - Centro Integral Oncológico Clara Campal Ensayos Clínicos START, Madrid
- Sweden (2):
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Karolinska Universitetssjukhuset, Solna
- United Kingdom (8):
  - Belfast City Hospital, Belfast
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Addenbrookes Hospital, Cambridge
  - Royal Liverpool University Hospital, Liverpool
  - Barts Health NHS Trust, London
  - Guys Hospital, London
  - Imperial College Healthcare NHS Trust - Hammersmith Hospital, London
  - University College London Cancer Institute, London

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing